CLINICAL TRIAL: NCT04555876
Title: High Tone External Muscle Stimulation On Endothelial Dysfunction And Walking Parameters In Peripheral Arterial Disease
Brief Title: Effect of High Tone External Muscle Stimulation on Peripheral Arterial Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rania Abdel Baset, principle invistigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: P.T.REC/012/002173
Record Dates: First submitted 2020-09-08; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Diabetic Peripheral Neuropathy

STUDY DESIGN:
Intervention Model Description: The patients will randomly be divided into two equal groups in number:
  1. Group A :
     Thirty patients will participate in physical therapy program in form of high-tone external muscle stimulation (HTEMS), with Frequencies continuously will be scanned from 4096 Hz to 31768 Hz, allowing for a much higher power of up to 5000 mW to be introduced 3 times per week, for 10 weeks plus supervised regular aerobic exercise program on stationary bicycle with moderate intensity, ( score 12-14 on Borg scale for rate of perceived exertion) 40 minutes per session, 3 times per week, for 10 weeks .
  2. Group B:
  Thirty patients will participate in a supervised regular aerobic exercise program only on stationary bicycle with moderate intensity, (score 12-14 on Borg scale for rate of perceived exertion) 40 minutes per session, 3 times per week, for 10 weeks.
Who Masked: Participant
Masking Description: The patients will randomly be divided into two equal groups in number:
  1. Group A :
     Thirty patients will participate in physical therapy program in form of high-tone external muscle stimulation (HTEMS), with Frequencies continuously will be scanned from 4096 Hz to 31768 Hz, allowing for a much higher power of up to 5000 mW to be introduced 3 times per week, for 10 weeks plus supervised regular aerobic exercise program on stationary bicycle with moderate intensity, ( score 12-14 on Borg scale for rate of perceived exertion) 40 minutes per session, 3 times per week, for 10 weeks .
  2. Group B:
  Thirty patients will participate in a supervised regular aerobic exercise program only on stationary bicycle with moderate intensity, (score 12-14 on Borg scale for rate of perceived exertion) 40 minutes per session, 3 times per week, for 10 weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high tone external muscle stimulation (Experimental): - HiTop 191 appliance (gbo Medizintechnik AG, Rimbach, Germany) Device HiToP® 4 touch gbo Medizintechnik AG, this modern high-tech design with brushed aluminum surface and the 15" TFT LC D full color touch screen monitor offer to the health care professional an indispensable feature.
  Interventions: Device: high tone external muscle stimulation- stationary bicycle
- stationary bicycle (Experimental): supervised regular aerobic exercise program on stationary bicycle with moderate intensity, (score 12-14 on Borg scale for rate of perceived exertion) 40 minutes per session, 3 times per week, for 10 weeks.
  Interventions: Device: high tone external muscle stimulation- stationary bicycle

INTERVENTIONS:
Device: high tone external muscle stimulation- stationary bicycle — high-tone external muscle stimulation (HTEMS), with Frequencies continuously will be scanned from 4096 Hz to 31768 Hz, allowing for a much higher power of up to 5000 mW to be introduced 3 times per week, for 10 weeks
  Other Names: stationary bicycle

SUMMARY:
to investigate the effect of high tone external muscle stimulation (HTEMS) on endothelial dysfunction and walking parameters in peripheral vascular disease.

DETAILED DESCRIPTION:
The patients will randomly be divided into two equal groups in number:

1. Group A :

   Thirty patients will participate in physical therapy program in form of high-tone external muscle stimulation (HTEMS), with Frequencies continuously will be scanned from 4096 Hz to 31768 Hz, allowing for a much higher power of up to 5000 mW to be introduced 3 times per week, for 10 weeks plus supervised regular aerobic exercise program on stationary bicycle with moderate intensity, ( score 12-14 on Borg scale for rate of perceived exertion) 40 minutes per session, 3 times per week, for 10 weeks .
2. Group B:

Thirty patients will participate in a supervised regular aerobic exercise program only on stationary bicycle with moderate intensity, (score 12-14 on Borg scale for rate of perceived exertion) 40 minutes per session, 3 times per week, for 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 1- Both genders are allowed to participate in the study. 2- The age range of patients will be from 50-60 years 3- All patients are diabetic from 5-7 years. 4- ABPI for all patients will be ranged from 0.65 to 0. 9 5- All patients are medically and psychologically stable. 6- Only ambulant patient without any aids will be selected 7- All patients are non smokers.

Exclusion Criteria:

1. Patients with ABPI ( Ankle Brachial Pressure Index ≤ 0.4 )
2. Patients who are unable to walk on treadmill or unable to attend sessions at the physical therapy department at Cairo university hospitals, 3 times a week.
3. Patients with unstable cardiovascular conditions (those with a known history of recent myocardial infarction, uncontrolled hypertension, ischemic attacks, stroke, and congestive heart failure) will be excluded from this study.
4. Patients with neurological problems that cause leg pain and polyneuropathy.
5. Patients with active malignancy will be excluded from study
6. Patients with ischemic ulcers or gangrenes
7. Patients with a vascular surgical procedure or angioplasty within the previous year will be excluded from the study
8. Patients with musculoskeletal disorders (Diagnosed with severe osteoporosis, severe osteoarthritis or joint replacement).

   -

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
measuring walking time in minutes | 10 weeks
  maximum walking time the patient can walk in minutes without complain
measuring walking distance in meter | 10 weeks
  maximum walking distance the patient can walk in meter

SECONDARY OUTCOMES:
Measuring serum Nitric Oxide | 10 weeks
  Three millimeter of venous blood will be drawn from the anticubital vein of each patient before conduction and after completion of the study. Blood sample will be drawn for Nitric Oxide (NO) measurement.